CLINICAL TRIAL: NCT03348657
Title: Decreased Risk of Falls in Patients Attending Music Sessions on an Acute Geriatric Ward
Brief Title: Risk of Falls in Patients Attending Music Sessions on an Acute Geriatric Ward
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Shek Fung, Principal Investigator, McGill University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMHC # 14-31
Record Dates: First submitted 2017-11-13; First posted 2017-11-21 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Fall; Music; Aged

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music intervention Group (Other): Patients who participated to at least one music session provided by volunteers while being admitted to the geriatric assessment unit. Participation to the music sessions was voluntary.
  Interventions: Other: Music Session
- Control Group (No Intervention): Patients who did not want to participate to the music sessions provided by volunteers while being admitted to the geriatric assessment unit

INTERVENTIONS:
Other: Music Session — Three to four times a week, volunteer musicians came to the geriatric assessment unit and would provide music sessions (duration of about 60 minutes) to the patients who volunteered to attend.
  Arms: Music intervention Group

SUMMARY:
Music therapy has long been used to improve communication, health and quality of life. Music is also known to regulate pain, mood and anxiety levels. In the geriatric population, music listening has been shown to decrease depressive symptoms and neuropsychiatric symptoms such as agitation and anxiety. As a result, the use of music is recommended by national guidelines to control the behavioural symptoms of patients in long-term care facilities. Despite the demonstrated positive benefits of music for health and behavioural outcomes, very few studies using music have been performed in the hospital environment and even fewer on short-stay geriatric units.

Older adults are the fastest-growing group of patients admitted to hospital, and the age-related burden of non-fatal health outcomes is one of the main challenges faced by hospitals. One of those age-related burdens is related to falls. Falls are highly frequent in geriatric patients, particularly on short-stay geriatric units, with a prevalence of up to 30 %. Falls are associated with increased length of hospital stay, high health-care costs and negative non-fatal health outcomes including multi-morbidities and related disabilities.

Previous research has shown that music may decrease the risk of falls. For example, it was shown that the rhythm of music, combined with physical exercise, can improve measures of gait stability. In older community dwellers, music-based programs have demonstrated that improvement of gait stability decreased the risk of falls. We therefore hypothesized that music listening may decrease the risk of falls of geriatric patients admitted to a short stay unit.

This study aimed to examine the influence of music listening on the risk of falls in patients admitted to a Geriatric Assessment Unit (GAU) by comparing the Morse Fall Scale (MFS) score for patients who attended music listening sessions and in control patients who did not attend these music sessions. To our knowledge, this is the first study to assess the effect of music listening on the risk of falls in a geriatric unit.

DETAILED DESCRIPTION:
Music is often used as a non-verbal means of emotional expression. As communication can be impaired in the elderly due to cognitive impairment and diseases, music can be used to recreate communication between the patients and their environment. Music therapy has long been used to improve communication, health and quality of life. Music is also known to regulate pain, mood and anxiety levels. In the geriatric population, music listening has been shown to decrease depressive symptoms and neuropsychiatric symptoms such as agitation and anxiety. As a result, the use of music is recommended by national guidelines to control the behavioural symptoms of patients in long-term care facilities. Despite the demonstrated positive benefits of music for health and behavioural outcomes, very few studies using music have been performed in the hospital environment and even fewer on short-stay geriatric units.

Older adults are the fastest-growing group of patients admitted to hospital, and the age-related burden of non-fatal health outcomes is one of the main challenges faced by hospitals. Thus, assessing and addressing the needs of the growing number of geriatric patients is necessary. One of those age-related burdens is related to falls. Falls are highly frequent in geriatric patients, particularly on short-stay geriatric units, with a prevalence of up to 30 %. Falls are associated with increased length of hospital stay, high health-care costs and negative non-fatal health outcomes including multi-morbidities and related disabilities.

Previous research has shown that music may decrease the risk of falls. For example, it was shown that the rhythm of music, combined with physical exercise, can improve measures of gait stability. In older community dwellers, music-based programs have demonstrated that improvement of gait stability decreased the risk of falls. We therefore hypothesized that music listening may decrease the risk of falls of geriatric patients admitted to a short stay unit.

This study aimed to examine the influence of music listening on the risk of falls in patients admitted to a Geriatric Assessment Unit (GAU) by comparing the Morse Fall Scale (MFS) score for patients who attended music listening sessions and in control patients who did not attend these music sessions. To our knowledge, this is the first study to assess the effect of music listening on the risk of falls in a geriatric unit.

ELIGIBILITY:
Inclusion Criteria:

* first admission to the GAU
* length of stay between 5 and 31 days

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Change in the risk of fall | At baseline (T0) and 4 weeks later (T1)
  The Morse Fall Scale (MFS). This is a rapid and simple method to assess the probability that a patient will fall. The total score is out of 125 and includes 6 items: history of previous falls, presence of a secondary diagnosis (i.e. more than one medical diagnosis in the patient's chart), use of an ambulatory aid (none, cane, walker), presence of intravenous therapy, gait and transfers (normal, weak, impaired) and the patient's mental status (oriented towards own ability or not). The score is further divided into 3 risk levels: low risk (less than 25 points), medium risk (25-44 points) and high risk (more than 45 points).

CONTACTS AND LOCATIONS:
Locations (1):
- St. Mary's Hospital Center, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Chabot J, Beauchet O, Fung S, Peretz I. Decreased risk of falls in patients attending music sessions on an acute geriatric ward: results from a retrospective cohort study. BMC Complement Altern Med. 2019 Mar 28;19(1):76. doi: 10.1186/s12906-019-2484-x. PMID 30922356